CLINICAL TRIAL: NCT05596851
Title: PSMA Radio-Guided Lymph Node Dissection With Beta-Probe, in High-risk Prostate Cancer Patients.
Brief Title: Radio-guided Surgery With DROP-IN Beta Probe for 68Ga-PSMA, in High-risk Prostate Cancer Patients Eligible for Robotic-assisted Radical Prostatectomy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1703
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Positron Emission Tomography; PSMA
Keywords: PSMA; Radio-Guided Surgery; Radio Guided Surgery; Lymph Node Dissection; Prostate Cancer; PET; Positron Emission Tomography
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the diagnostic efficacy and the safety of the combined approach with β-probe and 68Ga-PSMA-11 PET/CT in the correct identification of lymph node metastases, in high-risk prostate cancer patients undergoing radical prostatectomy and pelvic lymph node dissection.

DETAILED DESCRIPTION:
Study Phase: Phase II

Primary Objective:

To evaluate the diagnostic accuracy of the combined approach with β-probe and 68Ga-PSMA-11 PET/CT in the correct identification of lymph node metastases, in high-risk prostate cancer patients undergoing radical prostatectomy and pelvic lymph node dissection. The histopathological analysis of the surgical specimens will be considered the standard of reference and diagnostic accuracy will be evaluated in terms of sensitivity and specificity.

Secondary Objectives:

* the identification of the most appropriate tumor-to-background ratio (TBR) able to correctly locate the signal emitted by PSMA-positive lymph nodes compared with the signal derived by the background rumor.
* safety and toxicity analysis regarding the intraoperative application of the β-probe.
* the comparison between the signal detected by the β-probe and 68Ga-PSMA-11 PET/CT images.
* the correlation of the signal detected by the β-probe with the PSMA expression (PSMA staining) in lymph node metastases assessed by immuno-histochemical analysis on the surgical specimens

Drug Dosage, Formulation, Administration: Intravenous administration of 1.1 MBq/Kg of 68Ga-PSMA-11.

Primary Endpoint: Primary: sensitivity and specificity in a per-region analysis.

Secondary Endpoints:

* comparison of β-probe intra-operatory measurements with ex-vivo ones.
* comparison of β-probe measurements and 68Ga-PSMA-11 semi-quantitative parameters (SUVmax and PSMA-TV).
* comparison of β-probe measurements and PSMA expression assessed by IHC (PSMA staining).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer
* High-risk prostate cancer (T>T2c and/or PSA>20 and/or ISUP>3)
* Patients suitable for radical prostatectomy + pelvic lymph node dissection
* 68Ga-PSMA-11 PET/CT performed within 4 weeks prior to surgery
* PSMA positive pelvic lymph nodes detected at 68Ga-PSMA-11 PET/CT
* Age >18 years old
* Willing to sign informed consent

Exclusion Criteria:

* Patient unfit for surgery
* M1 stage (any M) detected at 68Ga-PSMA-11 PET/CT or other imaging modalities performed during diagnostic wok-up evaluation
* Unable to tolerate PET scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biopsy proven high-risk prostate cancer patients, who performed PSMA PET/CT per clinical routine practice will be considered suitable for enrollment in case of pelvic nodal involvement detected at PSMA PET/CT. Patients affected by metastatic prostate cancer (any M) will be considered not eligible.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and positive predictive value in a per-region analysis | March 2022 - March 2023

SECONDARY OUTCOMES:
Comparison of β-probe intra-operatory measurements with ex-vivo ones. | March 2022 - March 2023
Comparison of β-probe measurements and 68Ga-PSMA-11 semi-quantitative parameters | March 2022 - March 2023
  SUVmax and PSMA-TV will be evaluated as semi-quantitative parameters
Comparison of β-probe measurements and PSMA expression assessed by immunohistochemical analysis (IHC). | May 2022 - December 2023
  IHC will be evaluated by PSMA staining on the surgical specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- IEO European Institute of Oncology, Milan, Italy

REFERENCES:
- See also: IEO Nuclear Medicine — https://www.ieo.it/it/CHI-SIAMO/Come-siamo-organizzati/Le-divisioni/Divisione-di-Medicina-Nucleare-MNUDV/
- See also: Related Info — https://www.ieo.it/it/CHI-SIAMO/Come-siamo-organizzati/Le-divisioni/Divisione-di-Urologia-URODV/